CLINICAL TRIAL: NCT02817945
Title: 68Ga-NOTA-3P-TATE-RGD for Dual Somatostatin Receptor and Integrin αvβ3 PET/CT Imaging of Lung Cancer and Neuroendocrine Neoplams
Brief Title: Dual SSTR2 and Integrin αvβ3 Targeting PET/CT Imaging
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHNM13
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Lung Cancer; Neuroendocrine Neoplasm
Keywords: TATE-RGD; SSTR2; integrin αvβ3
MeSH Terms: conditions — Lung Neoplasms; Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-NOTA-3P-TATE-RGD PET/CT (Experimental): The patients were injected with 111-185 MBq of 68Ga-NOTA-3P-TATE-RGD in one dose intravenously and underwent PET/CT scan 45-60 min later.
  Interventions: Drug: 68Ga-NOTA-3P-TATE-RGD

INTERVENTIONS:
Drug: 68Ga-NOTA-3P-TATE-RGD — 68Ga-NOTA-3P-TATE-RGD were injected into the patients before the PET/CT scans

SUMMARY:
This is an open-label positron emission tomography/computed tomography (PET/CT) study to investigate the diagnostic performance and evaluate the efficacy of 68Ga-NOTA-3PTATE-RGD in lung cancer patients and neuroendocrine neoplam patients. A single dose of 111-185 Mega-Becquerel (MBq) 68Ga-NOTA-3P-TATE-RGD will be injected intravenously. Visual and semiquantitative method will be used to assess the PET/CT images.

DETAILED DESCRIPTION:
The number of somatostatin receptors may be greatly up-regulated in the cells of a variety of tumor including carcinoids, gastrinomas, paragangliomas, small cell lung cancer and non-small cell lung cancer. Octreotide is an eight amino acid cyclic peptide that preserves a four amino acid motif (Phe-Trp-Lys-Thr) that is critical for the biological activity of somatostatin (SSTR). On the other hand, the RGD moiety binds with integrin αvβ3, also plays an important role in the regulation of tumor growth, angiogenesis, local invasiveness, and metastatic potential in human tumor. To target both receptors, a heterodimeric peptide TATE-RGD was synthesized from TATE and RGD through a glutamate linker and then labeled with 68Ga. An open-label whole-body PET/ CT study was designed to investigate the safety and dosimetry of 68Ga-NOTA-3PTATE-RGD and diagnostic performance of 68Ga-NOTA-3PTATE-RGD PET/CT in evaluation of lung cancer and neuroendocrine neoplams.

ELIGIBILITY:
Inclusion Criteria:

* Neoplasm identified by X-ray, ultrasound or MRI as lung cancer or neuroendocrine tumors
* To provide basic information and sign the written informed consent.

Exclusion Criteria:

* Consisted of conditions of mental illness;
* Severe liver or kidney disease with serum creatinine > 3.0 mg/dl (270 μΜ) or any hepatic enzyme level 5 times or more than normal upper limit;
* Severe allergy or hypersensitivity to IV radiographic contrast
* Claustrophobia to accept the PET/CT scanning
* Pregnancy or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value of 68Ga-NOTA-3PTATE-RGD in lung cancer and Neuroendocrine Neoplasm | 1 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value (SUV) of the tracer in breast cancer will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospitall, Chinese Academy of Medical Science and Peking Union Medical College, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Jiang Y, Liu Q, Wang G, Sui H, Wang R, Wang J, Zhu Z. A prospective head-to-head comparison of 68 Ga-NOTA-3P-TATE-RGD and 68 Ga-DOTATATE in patients with gastroenteropancreatic neuroendocrine tumours. Eur J Nucl Med Mol Imaging. 2022 Oct;49(12):4218-4227. doi: 10.1007/s00259-022-05852-3. Epub 2022 Jun 3. PMID 35657429